CLINICAL TRIAL: NCT06356324
Title: The Effects of Music and Television on Intraoperative Hypertensive Events in Cataract Surgery: A Randomized Clinical Trial
Brief Title: The Effects of Music and Television on Intraoperative Hypertensive Events in Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021-13347
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Anxiety; Intraoperative Hypertension; Cataract
MeSH Terms: conditions — Anxiety Disorders; Cataract

STUDY DESIGN:
Intervention Model Description: Participants assigned to one of three groups: music listening, tv viewing, or control (waiting with ambient noise)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music intervention (Experimental): Participants instructed to listen to 20 minutes of relaxing classical music (e.g., Chopin, Mozart)
  Interventions: Other: Music Intervention
- Television intervention (Experimental): Participants instructed to watch a 20 minute segment of a relaxing home improvement show (e.g., House Hunters)
  Interventions: Other: Television Intervention
- Control (No Intervention): Participants instructed to wait in their preoperative room with no added stimulus intervention (i.e., music or television)

INTERVENTIONS:
Other: Music Intervention — Participants assigned to 20 minutes of music listening
  Arms: Music intervention
Other: Television Intervention — Participants assigned to 20 minutes of television viewing
  Arms: Television intervention

SUMMARY:
This study investigates whether television viewing or music listening can reduce pre-operative anxiety and improve surgical outcomes for patients undergoing cataract surgery. It aims to determine the effectiveness of these interventions compared to a control group and assess their impact on physiological markers of anxiety as well as the incidence of intra-operative hypertensive events.

The key questions that are to be answered are:

1. Does watching television before cataract surgery decrease intraoperative hypertensive events and/or pre-operative anxiety in patients?
2. Does listening to music before cataract surgery decrease intraoperative hypertensive events and/or pre-operative anxiety in patients?

DETAILED DESCRIPTION:
The study addresses the gap in literature regarding TV viewing's efficacy in ophthalmic surgery anxiety reduction. It aims to provide insights into cost-effective methods for stress reduction and surgical optimization. Through voluntary participation and rigorous methodology, it seeks to enhance patient experience and outcomes in ophthalmic surgery.

* Study Design: Randomized controlled design with three groups: control, television intervention, or music intervention.
* Objective: Investigate effects of TV viewing and music listening on pre-operative anxiety in ophthalmic surgery.
* Comparison: Compare relaxation effects of TV and music.
* Participants: Aim to recruit 200 per intervention arm from Montefiore Medical Center.
* Baseline Assessment: Measure anxiety levels pre-intervention.
* Interventions: Administer TV or music for 20 minutes pre-surgery.
* Assessment: Evaluate anxiety levels and physiological markers pre- and post-intervention.
* Monitoring: Monitor vital signs during surgery and post-operative period.
* Data Collection: Document demographic info, medical history, and baseline anxiety.
* Measurement Tools: Use Visual Analog Scale (VAS) for subjective assessment and physiological markers.
* Analysis: Compare outcomes across intervention arms using statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Participants undergoing cataract surgery at Montefiore Medical Center

Exclusion Criteria:

* Participants with severe hearing loss or speech impairment
* Participants with vision loss greater than count fingers
* Participants with uncontrolled hypertension (defined as >160/>100 despite use of antihypertensive medication)
* Participants who do not have the capacity to provide consent or who require a surrogate to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative hypertensive event | From beginning of cataract surgery to the completion (approximately 15 minutes)
  The primary outcome of this study is the occurrence of one hypertensive event (defined as BP >160/>100) during the procedure (cataract surgery).

SECONDARY OUTCOMES:
Change in VAS-A measurements for Anxiety | From participant enrollment to after 20 minute intervention
  The Visual Analog Scale for Anxiety (VAS-A) will be used to assess anxiety. The VAS-A is a validated tool for evaluating preoperative anxiety. Visual anxiety analog scale is used to score patient's anxiety levels. The scale ranges from 0 to 10, where 0 represents not anxious and 10 represents extreme anxiety. Participants have baseline measurements of VAS-A scores before 20 minute intervention, and after 20 minute intervention.
Change in Heart Rate measurements for Anxiety | From participant enrollment to after 20 minute intervention
  A physiological marker of anxiety is increased heart rate. As such, participants' heart rates will be measured (as heart beats per minute, bpm) and included in the data analysis. Participants have baseline measurements of heart rate before 20 minute intervention, and after 20 minute intervention.
Change in Blood pressure measurements for Anxiety | From participant enrollment to after 20 minute intervention
  A physiological marker of anxiety is increased blood pressure. As such, participants' blood pressures will be measured (systolic and diastolic pressure in mmHg) and included in the data analysis. Participants have baseline measurements of blood pressure before 20 minute intervention, and after 20 minute intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Barmettler, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No